CLINICAL TRIAL: NCT01614132
Title: Multicenter Pilot-study for the Therapy of Medulloblastoma of Adults (NOA-07)
Brief Title: Multicenter Pilot-study for the Therapy of Medulloblastoma of Adults
Acronym: NOA-07
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Peter Hau, Head, Clinical Neurooncology, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOA-07
Record Dates: First submitted 2012-04-26; First posted 2012-06-07 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Medulloblastoma
Keywords: medulloblastoma; CNS; malignant neoplasm; NOA; neuroectodermal tumor; Vincristin; CCNU; Cisplatin
MeSH Terms: conditions — Medulloblastoma; Neoplasms; Neuroectodermal Tumors | interventions — Maintenance Chemotherapy; Vincristine; Cisplatin; Lomustine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vincristin, CCNU, cis-platin (Experimental): radiotherapy and concomitant chemotherapy (7 cycles of 7 days):
  * 2 mg/m2 vincristin i.v.
  * 55,0 Gy Posterior cranial fossa (M0)
  * 55,0 Gy Posterior cranial fossa / cerebral metastases + 49,6 Gy spinal metastases (M1-M3)
  maintenance chemotherapy (8 cycles of 42 days):
  * once at day 1 at each cycle: 70 mg/m2 cis-platin i.v. 75 mg/m2 CCNU oral 2 mg/m2 vincristin i.v.
  * once at day 8 and 15 at each cycle: 2 mg/m2 vincristin i.v.
  Interventions: Drug: maintenance chemotherapy (vincristin, cisplatin and CCNU); Radiation: Radiotherapy

INTERVENTIONS:
Drug: maintenance chemotherapy (vincristin, cisplatin and CCNU) — maintenance chemotherapy of maximum of 8 cycles á 42 days
  Other Names: Vincristin: L01CA02; CCNU: Lomustin L01AD02; cis-platin: L01XA01
Radiation: Radiotherapy — Radiotherapy of the partial brain

SUMMARY:
The purpose of this study is to determine whether a combination of a radiochemotherapy (vincristin) and a following maintenance chemotherapy (vincristin, cisplatin and CCNU) in adult patients with medulloblastoma is tolerable.

DETAILED DESCRIPTION:
As medulloblastoma in adult patients are very rare (1.1% of all brain tumors), adults are often treated in the scope of expanded access treatments or within pediatric studies; although, it is not known whether medulloblastomas act in the same way in adulthood and in childhood. This is the first study to investigate the significance of a combination of a radiochemotherapy (vincristin) and a following maintenance chemotherapy (vincristin, cisplatin and CCNU) in adult patients with medulloblastoma with the purpose to have a starting point for the development of chemotherapeutical protocols in adults.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* medulloblastoma (+/- postoperative residual tumor, M0) or medulloblastoma (+/- postoperative residual tumor, M1-M3) respectively
* primary diagnosis of the tumor
* no previous chemo- or radiation therapy
* Karnofsky-Index ≥ 70%
* WBC ≥ 3000/μl; thrombocytes ≥ 100 000/μl; Hb ≥ 10 g/dl
* creatinine =< 1,5 ULN; Bilirubin =< 1,5 ULN; GPT, GOT, AP =< 2,5 ULN
* HIV and hepatitis B/C negative
* no factors / any medical condition affecting patient's compliance
* patient needs to fulfil protocol's requirements
* patient is willing to use highly effective methods of contraception during dosing and for 6 months after the last dose; women of child-bearing potential must have a negative hCG laboratory test at baseline; pregnancy tests must be repeated every 4 weeks
* patient's written consent

Exclusion Criteria:

* age < 18 years
* histologically not confirmed Medulloblastoma
* by chemo- or radiotherapy treated recidive tumor
* other cancer (with exception of surgically cured carcinoma in situ of the cervix and non-melanocytic skin tumors)
* hypersensitivity or contraindication against one of the used drugs
* current or planned participation to another clinical trial during this study Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrolment or could interfere with the patient participating in and completing the study
* Any medical condition associated with high medical risk or contraindicated to use chemotherapeutic agents as indicated in current product package insert
* Pregnant or nursing (lactating) women; women or men not willing to use a highly effective methods of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
feasibility of the adjuvant chemotherapy | participants will be followed for the duration of chemo therapy, an expected average of 1 year
  The main objective is the feasibility of the adjuvant chemotherapy which has gained the best results when combined with radiotherapy so far.
  The present protocol is primarily to determine the number of interruptions of the maintenance chemotherapy due to toxicity and the kind of toxicity .

SECONDARY OUTCOMES:
Number of performable cycles in chemo therapy | participants will be followed for the duration of chemo therapy, an expected average of 6 months
  It should be determined how many cycles in the maintenance chemotherapy are feasible.
3 and 5 years progression-free survival | participants will be followed for the duration of chemo therapy and in the follow-up periode, an expected average of 3 to 5 years
  The 3 and 5-years rate of progression-free survival (pfs) should be determined for adult patients.
event-free survival | participants will be followed for the duration of chemo therapy and in the follow-up periode, an expected average of 3 to 5 years
  The event-free survival (efs) should be determined for adult patients.
overall survival | participants will be followed for the duration of chemo therapy and in the follow-up periode, an expected average of 3 to 5 years
  The overall survival (os) should be determined for adult patients.
course of cognitive performance/QoL | participants will be followed for the duration of chemo therapy and in the follow-up periode, an expected average of 3 to 5 years
  The course of the cognitive performance and the quality of life should be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hau, MD, Principal Investigator — Department of Neurology, University of Regensburg
Locations (15):
- Germany (15):
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Neurologische Universitätsklinik, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Otto-von-Guericke Universität, Magdeburg
  - Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Katharinenhospital, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided